CLINICAL TRIAL: NCT03784001
Title: Cultivating Gratitude: Does Manipulating Expectations Improve the Efficacy of a Gratitude Intervention?
Brief Title: The Effects of Manipulating Expectations in a Gratitude Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Tanera van Diggelen, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1997
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Gratitude + No Expectations; Gratitude + Expectations; Events Control
Keywords: Gratitude, Expectations, Well-being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three conditions: Gratitude, Gratitude + Expectations, or Events Control Participants in the two gratitude conditions will login to an online Google form three times a week for two weeks and make entries of up to five things they are grateful for. The form for participants in the gratitude + expectation condition will also provide information about benefits of gratitude. An everyday events control will be used to provide a neutral comparison condition. This group will be instructed to type up to five things or events of note from their day on their form.
Who Masked: Participant
Masking Description: Participants will only know they are taking part in a "Mood and Writing Study" and will not know which condition they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gratitude + No Expectations (Active Comparator): Participants will type online lists of up to five items they are grateful for, every two days for two weeks.
  Interventions: Behavioral: Gratitude + No Expectations Intervention
- Gratitude + Expectations (Experimental): Participants will type online lists of up to five items they are grateful for, every two days for two weeks. They will also be told a benefit of gratitude each time they write an online gratitude list.
  Interventions: Behavioral: Gratitude + Expectations Intervention
- Events Control (Active Comparator): Participants will type online lists of up to five events from their day, every two day for two weeks.
  Interventions: Behavioral: Events Control Intervention

INTERVENTIONS:
Behavioral: Gratitude + No Expectations Intervention — Participants will be emailed six different times, once every two days, with a link to an anonymous Google form. Each Google form will instruct participants to type a short gratitude list of up to five items. Additionally, the first form will include a demographics questionnaire and the first and sixth forms will include questionnaires assessing all outcomes of interest
  Arms: Gratitude + No Expectations
Behavioral: Gratitude + Expectations Intervention — Participants will be emailed six different times, once every two days, with a link to an anonymous Google form. Each Google form will instruct participants to type a short gratitude list of up to five items. Participants will have a statement at the top of their Google form about the benefits of gratitude. Examples of these statements are: "Practicing gratitude may increase social connectedness" and "Cultivating gratitude was shown to improve school satisfaction in a UK sample of students". Additionally, the first form will include a demographics questionnaire and the first and sixth forms will include questionnaires assessing all outcomes of interest
  Arms: Gratitude + Expectations
Behavioral: Events Control Intervention — Participants will be emailed six different times, once every two days, with a link to an anonymous Google form. Each Google form will instruct participants to type a list of up to five items about events from their day. Additionally, the first form will include a demographics questionnaire and the first and sixth forms will include questionnaires assessing all outcomes of interest.
  Arms: Events Control

SUMMARY:
Gratitude - an emotion felt when an individual receives something beneficial from other people or entities - has been shown to positively affect well-being. Beginning in 2003, "count your blessings" interventions - in which participants list items they are grateful for, and gratitude letter writing interventions were designed to cultivate gratitude. Gratitude interventions have many positive outcomes; they can increase well-being and life satisfaction (Froh, Sefick, & Emmons, 2008) and increase self-esteem (Rash, Matsuba, & Prkachin, 2011) to name a few.

Knowing the benefits of gratitude prior to an intervention could affect participant behavior and health outcomes. Past studies have illustrated that sharing information about treatments changes expectations and improves outcomes (Zion & Crum, 2018). For instance, overt medical treatments are more effective than hidden ones (Colloca, Lopiano, Lanotte, & Benedetti, 2004).

The proposed study is designed to evaluate whether expectations about intervention efficacy can enhance the benefits of a brief gratitude intervention. Specifically, the investigators will test if providing information on the benefits of gratitude will enhance intervention outcomes. This 3-armed randomized controlled trial will have the following conditions: gratitude + expectation, gratitude, and events control. Participants will be undergraduate college students and the online intervention will last two weeks.

Participants in the two gratitude conditions will login to an online form three times a week for two weeks and make entries of up to five things they are grateful for. The form for participants in the gratitude + expectation condition will also provide information about benefits of gratitude. An everyday events control will be used to provide a neutral comparison condition. This group will be instructed to type up to five things or events of note from their day on their form.

Outcome measures will be collected via an online survey before and immediately after the intervention. The primary outcome is well-being and the secondary outcomes are sleep quality and quantity, state gratitude, positive affect, healthcare self-efficacy, stress, and depressive symptoms. The investigators predict that participants in the gratitude + expectation condition will have enhanced intervention outcomes compared to participants in comparison conditions.

DETAILED DESCRIPTION:
Overview: Potential participants will be recruited from an undergraduate psychology class. Participants will have one week after initial study advertisement to read the consent form and decide if they wish to participate. When participants turn in a signed consent form, they will be officially enrolled in the study and issued a personal identification (PI) number to use throughout the study.

Participants will be randomly assigned to one of three conditions: gratitude + expectations, gratitude, or an everyday events control condition. Participants will be emailed six different times, once every two days, with a link to an anonymous Google form. Each Google form will instruct participants to type either a short gratitude list (for gratitude + expectations and gratitude conditions) or an events list (for everyday events control), and will have a section for participants to enter their personal identification numbers. Additionally, the first form will include a demographics questionnaire and the first and sixth forms will include questionnaires assessing all outcomes of interest.The primary outcome of interest is well-being. The secondary outcomes of interest are sleep, state gratitude, healthcare self-efficacy, stress, and depressive symptoms.

Participants in the gratitude + expectations condition will have a statement at the top of their Google form about the benefits of gratitude. Examples of these statements are: "Practicing gratitude may increase social connectedness" and "Cultivating gratitude was shown to improve school satisfaction in a sample of students". By the end of the study, participants will have completed six gratitude or everyday events lists and two questionnaires.

Interventions:

1. Gratitude + No Expectations: Participants in the gratitude condition will practice a counting your blessings intervention for two weeks. Participants will be instructed to list up to five things they are grateful for every two days for the two weeks of the intervention (six times total).
2. Gratitude + expectations: Participants in this condition will be given the same instructions as the gratitude condition and will also be given the regular reminders of the benefits of gratitude.
3. Everyday events: Participants will be instructed to list up to five details about their day, such as activities they engaged in, or conversations they had. Participants will make these lists every two days for two weeks (six times total).

Questionnaires:

Self-report questionnaires with high test-retest reliability and internal validity will be administered at baseline and post intervention to access changes in outcomes of interest, such as well-being, depressive symptoms, and anxiety.

Questionnaires administered only at baseline: Communication and Attitudinal Self-Efficacy Scale (CASE) and demographic questionnaire

Questionnaires administered pre- and post-intervention: Mental Health Continuum-Short Form, Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Scale, Pittsburg Sleep Quality Index (PSQI) duration items, Modified Differential Emotions Scale, Center for Epidemiologic Studies Depression Scale (CES-D), Perceived Stress Scale 4

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate Student
* Proficient in English
* 18 years of age or older
* Has a valid email address
* Access to the internet

Exclusion Criteria:

-No other exclusion criteria (aside from meeting the inclusion criteria above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanera van Diggelen, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Froh JJ, Sefick WJ, Emmons RA. Counting blessings in early adolescents: an experimental study of gratitude and subjective well-being. J Sch Psychol. 2008 Apr;46(2):213-33. doi: 10.1016/j.jsp.2007.03.005. Epub 2007 May 4. PMID 19083358
- [Background] Bartlett MY, DeSteno D. Gratitude and prosocial behavior: helping when it costs you. Psychol Sci. 2006 Apr;17(4):319-25. doi: 10.1111/j.1467-9280.2006.01705.x. PMID 16623689
- [Background] Watkins, P., Woodward, K., Stone, T., & Kolts, R. (2003). Gratitude and happiness: Development of a measure of gratitude and relationships with subjective well-being. Social Behavior and Personality: An international journal, 31, 431-452. doi: 10.2224/sbp.2003.31.5.431
- [Background] Kruse, E., Chancellor, J., Ruberton, P.M., & Lyubomirsky, S. (2014). An upward spiral between gratitude and humility. Social Psychological and Personality Science. 5(7), 805-814. doi: 10.1177/1948550614534700
- [Background] Rash, J. A., Matsuba, M. K., & Prkachin, K. M. (2011). Gratitude and well-being: who benefits the most from a gratitude intervention? Applied Psychology: Health and Well-Being, 3(3), 350-369. doi: 10.1111/j.1758-0854.2011.01058.x
- [Background] Zion SR, Crum AJ. Mindsets Matter: A New Framework for Harnessing the Placebo Effect in Modern Medicine. Int Rev Neurobiol. 2018;138:137-160. doi: 10.1016/bs.irn.2018.02.002. Epub 2018 Mar 20. PMID 29681322
- [Background] Colloca L, Lopiano L, Lanotte M, Benedetti F. Overt versus covert treatment for pain, anxiety, and Parkinson's disease. Lancet Neurol. 2004 Nov;3(11):679-84. doi: 10.1016/S1474-4422(04)00908-1. PMID 15488461
- [Background] Emmons RA, McCullough ME. Counting blessings versus burdens: an experimental investigation of gratitude and subjective well-being in daily life. J Pers Soc Psychol. 2003 Feb;84(2):377-89. doi: 10.1037//0022-3514.84.2.377. PMID 12585811
- [Background] Sheldon, K.M. & Lyubomirsky, S. 2006. How to increase and sustain positive emotion: The effects of expressing gratitude and visualizing best possible selves. The Journal of Positive Psychology. 1(2). 73-82. doi:10.1080/17439760500510676
- [Background] Jackowska M, Brown J, Ronaldson A, Steptoe A. The impact of a brief gratitude intervention on subjective well-being, biology and sleep. J Health Psychol. 2016 Oct;21(10):2207-17. doi: 10.1177/1359105315572455. Epub 2015 Mar 2. PMID 25736389

RESULTS

PARTICIPANT FLOW:
Groups:
- Gratitude + No Expectations (GNE): Participants will type online lists of up to five items they are grateful for, every two days for 13 days.
  Gratitude Intervention: Participants will be emailed six different times, once every two days, with a link to an anonymous Google form. Each Google form will instruct participants to type a short gratitude list of up to five items.
- Gratitude + Expectation (GE): Participants will type online lists of up to five items they are grateful for, every two days for 13 days. They will also be told a benefit of gratitude each time they write an online gratitude list.
  Gratitude + Expectations Intervention: Participants will be emailed six different times, once every two days, with a link to an anonymous Google form. Each Google form will instruct participants to type a short gratitude list of up to five items. Participants will have a statement at the top of their Google form about the benefits of gratitude. Examples of these statements are: "Practicing gratitude may increase social connectedness" and "Cultivating gratitude was shown to improve school satisfaction in a UK sample of students".
- Events Control: Participants will type online lists of up to five events from their day, every two day for 13 days.
  Events Control Intervention: Participants will be emailed six different times, once every two days, with a link to an anonymous Google form. Each Google form will instruct participants to type a list of up to five items about events from their day.
Period: Overall Study
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Started (The number of participants who completed their baseline questionnaire and first list.) | 46 | 38 | 41
Completed | 44 | 38 | 40
Not Completed | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control | Total
Number analyzed (Participants) | 46 | 38 | 41 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.46 (2.43) | 22.00 (3.30) | 21.27 (1.18) | 21.56 (2.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 28 | 30 | 96
  Male | 8 | 10 | 11 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/ Caucasian | 23 | 9 | 13 | 45
  Hispanic/ Latino/a | 9 | 7 | 5 | 21
  Asian | 10 | 14 | 18 | 42
  Native Hawaiian, American Indian or Alaska Native | 3 | 6 | 2 | 11
  Black or African American | 1 | 2 | 3 | 6
School Year (4th Year of Undergraduate Study) [Count of Participants; unit: Participants] | 33 | 29 | 28 | 90
Family Income, Categorical (> $100,000/ year) [Count of Participants; unit: Participants] | 22 | 14 | 20 | 56

OUTCOME MEASURES:

1. Primary Outcome: Mental Health Continuum-Short Form (MHC-SF)
Description: Hedonic well-being, eudaimonic well-being, and overall well-being were assessed at baseline and post-intervention. Well-being was measured with the Mental Health Continuum-Short Form (MHC-SF; Keyes, 2009). Participants rated how often they felt 14 different emotions or statements, such as "happy" and "satisfied with life". Items are rated on a 6-point likert scale (0 = never, 5 = everyday). This measure assesses both hedonic and eudaimonic well-being. The MHC-SF is both reliable and valid for use with young adults (Robitschek & Keyes, 2009). Total scores are created by the sum of scores for all 14 items, with a range of 0-70. Higher scores indicate greater overall well-being.
Time Frame: Assessed at Pre- and Post- Intervention (2 weeks apart)
Population: These are the numbers analyzed when assessing overall well-being
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Number analyzed (Participants) | 41 | 38 | 38
score on a scale
  Pre-Intervention | 26.15 (7.512) | 21.29 (8.60) | 24.37 (9.35)
  Post-intervention | 26.78 (7.82) | 23.21 (9.19) | 23.95 (10.21)

2. Primary Outcome: Mental Health Continuum-Short Form (MHC-SF): Hedonic Well-Being SubScale
Description: Well-being was measured with the Mental Health Continuum-Short Form (MHC-SF; Keyes, 2009). Participants rated how often they felt 14 different emotions or statements, such as "happy" and "satisfied with life". Items are rated on a 6-point likert scale (0 = never, 5 = everyday), with higher numbers indicating greater well-being. This measure assesses both hedonic and eudaimonic well-being. The MHC-SF is both reliable and valid for use with young adults (Robitschek & Keyes, 2009). The Hedonic Well-Being Subscale is the sum of items 1-3 on the Mental Health Continuum Short-Form. Total scores range from 0-15, with higher scores indicating greater hedonic well-being. Scoring a 4 or 5 on at least one of the 3 items on the Hedonic Well-Being Subscale indicates a diagnosis of flourishing mental health.
Time Frame: Assessed at Pre- and Post- Intervention (2 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Number analyzed (Participants) | 42 | 38 | 38
score on a scale
  Pre-Intervention | 5.86 (1.84) | 4.95 (2.36) | 5.84 (1.84)
  Post-intervention | 6.24 (1.79) | 5.03 (2.50) | 5.39 (2.56)

3. Primary Outcome: Mental Health Continuum-Short Form (MHC-SF): Eudaimonic Well-Being SubScale
Description: Well-being was measured with the Mental Health Continuum-Short Form (MHC-SF; Keyes, 2009). Participants rated how often they felt 14 different emotions or statements, such as "happy" and "satisfied with life". Items are rated on a 6-point likert scale (0 = never, 5 = everyday), with higher numbers indicating greater well-being. This measure assesses both hedonic and eudaimonic well-being. The MHC-SF is both reliable and valid for use with young adults (Robitschek & Keyes, 2009). The score of the Eudaimonic Subscale is the sum of items 4-14 on the MHC-SF. Scores range from 0-55. Higher scores indicate greater eudaimonic well-being (i.e., greater social and psychological well-being).
Time Frame: Assessed at Pre- and Post- Intervention (2 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Number analyzed (Participants) | 42 | 38 | 38
score on a scale
  Pre-Intervention | 20.21 (5.94) | 16.34 (6.51) | 18.53 (7.53)
  Post-intervention | 20.52 (6.31) | 18.18 (7.02) | 18.55 (7.96)

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Scale
Description: Sleep quality was measured with the 8-item PROMIS sleep disturbance short form (Yu et al., 2012). Participants rated their level of agreement with eight different statements about their sleep in the past seven days such as "My sleep was restless" and "I had difficulty falling asleep". Participants rated each item on a 5 point scale (1 = not at all, 5 = very much). Items 2, 3, 7, and 8 were reverse scored. The total score of the PROMIS Sleep Disturbance Scale is the sum of the scores for all 8 items. Total scores range from 8-40, with higher scores indicating more severe sleep disturbance.
Time Frame: Assessed at Pre- and Post- Intervention (2 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Number analyzed (Participants) | 41 | 37 | 38
score on a scale
  Pre-Intervention | 21.05 (6.62) | 25.43 (7.08) | 20.71 (6.90)
  Post-intervention | 19.17 (7.52) | 23.38 (7.8) | 20.61 (6.98)

5. Secondary Outcome: Pittsburg Sleep Quality Index (PSQI) Duration Items
Description: Sleep quantity was measured with the Pittsburgh Sleep Quality Index Duration Items (PSQI-4), which asks participants questions such as when they went to bed and when they woke up in the morning (Buysse et al., 1989). PSQI duration items are questions 1-4 on the PSQI, which measure how much sleep respondents have been getting. Higher hours of sleep is a better outcome.
Time Frame: Assessed at Pre- and Post- Intervention (2 weeks apart)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Number analyzed (Participants) | 41 | 37 | 38
hours
  Pre-Intervention | 6.56 (1.42) | 5.91 (1.29) | 6.30 (1.09)
  Post-intervention | 6.86 (0.95) | 6.26 (1.60) | 6.68 (1.45)

6. Secondary Outcome: Modified Differential Emotions Scale (MDES): Positive Emotions Subscale
Description: Positive affect was measured with the ten-item Positive Emotions (PE) subscale of the Modified Differential Emotions Scale (mDES) (Fredrickson, Tugade, Waugh, and Larkin, 2003). Participants rated how often they felt ten different groups of positive emotions such as "amused, fun-loving, silly" on a 5-point scale (0 = not at all, 4 = most of the time). The average of the items was calculated to measure positive affect, with higher numbers indicating greater positive affect.
Time Frame: Assessed at Pre- and Post- Intervention (2 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Number analyzed (Participants) | 43 | 37 | 38
score on a scale
  Pre-Intervention | 2.86 (0.72) | 2.57 (0.80) | 2.78 (0.76)
  Post-intervention | 2.85 (0.80) | 2.71 (0.85) | 2.84 (0.84)

7. Secondary Outcome: Perceived Stress Scale - 4 (PSS-4)
Description: Stress was measured with the 4-item Perceived Stress Scale (PSS-4; Cohen, Kamarack, and Mermelstein, 1983). Participants rated how often they felt a certain way in the last week on four different items such as "How often have you felt confident about your ability to handle your personal problems?" and "How often have you felt that things were going your way?" on a 5- point scale (0 = never, 4 = very often). The total score of the PSS-4 is the sum of all 4 items. Total scores range from 0-16, and higher scores indicate greater perceived stress.
Time Frame: Assessed at Pre- and Post- Intervention (2 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Number analyzed (Participants) | 42 | 38 | 38
score on a scale
  Pre-Intervention | 7.05 (3.17) | 7.95 (3.17) | 6.03 (3.18)
  Post-intervention | 6.62 (3.22) | 6.89 (3.03) | 6.16 (3.33)

8. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D)
Description: Depressive symptoms were measured by the Center for Epidemiological Studies - Depression Scale (CES-D, Radloff, 1977). Participants rated how often they experienced 20 different statements such as "I was bothered by things that usually don't bother me" and "I felt like everything I did was an effort" in the past week. Participants scored each item on a 4-point scale (0 = rarely or none of the time 3 = all of the time). The total score for the CES-D is the sum of all 20 items, with a range of 0-60, with higher scores indicating greater depressive symptoms.
Time Frame: Assessed at Pre- and Post- Intervention (2 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Number analyzed (Participants) | 42 | 38 | 37
score on a scale
  Pre-Intervention | 17.21 (9.97) | 21.95 (13.12) | 17.08 (11.19)
  Post-intervention | 17.40 (12.45) | 18.47 (12.96) | 17.08 (12.96)

9. Secondary Outcome: Modified Differential Emotions Scale (MDES): State Gratitude
Description: State gratitude was measured with item one of the mDES (Fredrickson, Tugade, Waugh, and Larkin, 2003), which asks participants how often they felt "grateful, appreciative, or thankful" in the past two weeks. Participants rated this item on a 5-point scale (0 = not at all, 4 = most of the time), with a higher number indicating higher feelings of gratitude.
Time Frame: Assessed at Pre- and Post- Intervention (2 weeks apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
Number analyzed (Participants) | 43 | 37 | 38
score on a scale
  Pre-Intervention | 3.07 (0.74) | 2.95 (0.98) | 3.11 (0.83)
  Post-intervention | 3.05 (0.84) | 3.05 (0.91) | 3.13 (0.91)

ADVERSE EVENTS:
Time Frame: Because this was a short behavioral study of minimal risk to participants, we did not monitor for adverse events. We let participants know that they could drop out of the study at any time and could choose not to answer any questions that they would not like to answer on the questionnaires.
Description: Because this was a short behavioral study of minimal risk to participants, we did not monitor for adverse events. We let participants know that they could drop out of the study at any time and could choose not to answer any questions that they would not like to answer on the questionnaires.
Arm/Group | Gratitude + No Expectations (GNE) | Gratitude + Expectation (GE) | Events Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03784001/Prot_SAP_000.pdf